CLINICAL TRIAL: NCT05174507
Title: Empagliflozin and Anakinra for the Treatment of Postprandial Hypoglycemia in Patients With Prediabetes: a Randomized, Placebo-controlled Study
Brief Title: Empagliflozin and Anakinra for the Treatment of Postprandial Hypoglycemia in Patients With Prediabetes
Acronym: Hypo-PrEA
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: 2020-01287; me20Donath
Record Dates: First submitted 2021-12-13; First posted 2021-12-30 (Actual); Last update posted 2024-02-20 (Actual); Status verified 2024-02

CONDITIONS: Postprandial Hypoglycemia
Keywords: SGLT2-inhibitor empagliflozin; IL-1 receptor antagonist anakinra; prediabetes; insulin clearance; proinsulin
MeSH Terms: conditions — Hypoglycemia; Prediabetic State; Diabetes Mellitus, Insulin-Dependent, 2 | interventions — empagliflozin; Interleukin 1 Receptor Antagonist Protein

STUDY DESIGN:
Intervention Model Description: Placebo controlled, double-blind, randomized, cross-over proof-of-concept study. Subjects will be randomized to either group 1-6 (ratio 1:1, in blocks of 4 participants).
Who Masked: Participant, Care Provider, Investigator
Masking Description: Participants, investigators and study nurses will be blinded to the study drug.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Group 1 (anakinra; placebo; empagliflozin) (Other): Group 1:
  study day 1: anakinra; study day2: placebo; study day 3: empagliflozin
  Interventions: Drug: empagliflozin; Drug: anakinra; Other: saline subcutaneous (s.c.) (placebo); Other: tablet per oral (p.o.) (placebo)
- Group 2 (placebo; anakinra; empagliflozin) (Other): study day 1: placebo; study day2: anakinra; study day 3: empagliflozin
  Interventions: Drug: empagliflozin; Drug: anakinra; Other: saline subcutaneous (s.c.) (placebo); Other: tablet per oral (p.o.) (placebo)
- Group 3 (empagliflozin; placebo; anakinra) (Other): study day 1: empagliflozin; study day2: placebo; study day 3: anakinra
  Interventions: Drug: empagliflozin; Drug: anakinra; Other: saline subcutaneous (s.c.) (placebo); Other: tablet per oral (p.o.) (placebo)
- Group 4 (empagliflozin; anakinra; placebo) (Other): study day 1: empagliflozin; study day2: anakinra; study day 3: placebo
  Interventions: Drug: empagliflozin; Drug: anakinra; Other: saline subcutaneous (s.c.) (placebo); Other: tablet per oral (p.o.) (placebo)
- Group 5 (placebo; empagliflozin; anakinra) (Other): study day 1: placebo; study day2: empagliflozin; study day 3: anakinra
  Interventions: Drug: empagliflozin; Drug: anakinra; Other: saline subcutaneous (s.c.) (placebo); Other: tablet per oral (p.o.) (placebo)
- Group 6 (anakinra; empagliflozin; placebo) (Other): study day 1:anakinra; study day2: empagliflozin; study day 3: placebo
  Interventions: Drug: empagliflozin; Drug: anakinra; Other: saline subcutaneous (s.c.) (placebo); Other: tablet per oral (p.o.) (placebo)

INTERVENTIONS:
Drug: empagliflozin — Empagliflozin (Jardiance®; Boehringer Ingelheim (Schweiz) GmbH) is a highly selective, reversible inhibitor of the sodium glucose co-transporter 2 (SGLT2). Treatment consists of a single oral tablet of 25 mg of empagliflozin (Jardiance®) two hours before ingestion of the mixed-meal (Ensure plus® 375 ml, 75 g carbohydrates, 562 kcal, drinking time 5 minutes).
Drug: anakinra — Anakinra (Kineret®; r-metHuIL-1ra, Swedish Orphan Biovitrum AB) is a recombinant, non-glycosylated form of the human interleukin-1 receptor antagonist (IL-1Ra) in a 100 mg/0.67ml solution for SC injection. Treatment consists of a single subcutaneous injection of 100 mg Anakinra (Kineret®) three hours before ingestion of the mixed-meal (Ensure plus® 375 ml, 75 g carbohydrates, 562 kcal, drinking time 5 minutes).
Other: saline subcutaneous (s.c.) (placebo) — Placebo for anakinra is 0.67 ml of sterile 0.9 % saline solution s. c. Treatment consists of a single subcutaneous injection of matched placebo (0.67 ml of 0.9 % saline) three hours before ingestion of the mixed-meal (Ensure plus® 375 ml, 75 g carbohydrates, 562 kcal, drinking time 5 minutes).
Other: tablet per oral (p.o.) (placebo) — Placebo for empagliflozin is Winthrop P® (Zentiva, Frankfurt/Main) lactose tablet. Treatment consists of a single oral tablet of matched placebo two hours before ingestion of the mixed-meal (Ensure plus® 375 ml, 75 g carbohydrates, 562 kcal, drinking time 5 minutes).

SUMMARY:
This study is to analyze whether the SGLT2-inhibitor empagliflozin or the IL-1 receptor antagonist anakinra may improve postprandial hypoglycemia in subjects with prediabetes.

DETAILED DESCRIPTION:
Subjects with prediabetes may develop postprandial hypoglycemia. This is probably due to a dysfunction of the insulin producing β-cell characterized by a delayed and exaggerated insulin secretion leading to an initial peak in glycaemia followed by a rapid fall and eventually resulting in hypoglycemia. The latter occurring typically within 1 to 3 hours after food intake.

In patients with gastric bypass surgery and postprandial hypoglycemia the SGLT2-inhibitor empagliflozin and the IL-1 receptor antagonist anakinra reduced postprandial insulin release and prevented hypoglycemia. This study is to analyze whether a similar therapeutic approach using empagliflozin and anakinra may also improve postprandial hypoglycemia in subjects with prediabetes.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with prediabetes defined by Glycosylated haemoglobin A1c (HbA1c) 5.7-6.4 % or fasting plasma glucose 6.1-6.9 mmol/l) or plasma glucose 2 h following 75 glucose ingestion of 7.8-11.0 mmol/l.
* Hypoglycemia occuring 1 to 3 h following ingestion of a standardized liquid mixed-meal (75 g carbohydrates) and fulfilling the Whipple's triad (glucose below 3.0 mmol/l).
* Age ≥ 18 years
* For subjects with reproductive potential, willingness to use contraceptive measures adequate to prevent the subject from becoming pregnant during the study

Exclusion Criteria:

* Upper gastrointestinal surgery
* Diagnosis of any type of diabetes mellitus
* Signs of current infection
* Use of investigational drug up to one week prior to start of treatment phase
* Glucocorticoid therapy
* Neutropenia (leukocyte count < 1.5 × 109/L or absolute neutrophil count (ANC) < 0.5 × 109/L)
* Anemia (hemoglobin < 11 g/dL for males, < 10 g/dL for females)
* Clinically significant kidney or liver disease (creatinine > 1.5 mg/dL, aspartate aminotransferase (AST)/ALT > 2 × ULN, alkaline phosphatase > 2 × ULN, or total bilirubin [tBili] > 1.5 × ULN)
* Uncontrolled disease
* Currently pregnant or breastfeeding
* No subjects meeting the criteria for vulnerability
* Participation in another study with investigational drug within the 30 days preceding and during the present study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Estimated)
Dates: Start 2022-06-24 (Actual); Primary Completion 2024-05 (Estimated); Study Completion 2024-05 (Estimated)

PRIMARY OUTCOMES:
Number of symptomatic hypoglycemia | up to 3 hours after ingestion of the liquid mixed-meal
  Incidence of symptomatic hypoglycemia following a standardized mixed-meal test defined by appearance of typical symptoms, blood glucose level below 3.0 mmol/l and relief of symptoms when the glucose level is raised (Whipple's triad).

SECONDARY OUTCOMES:
Severity of symptoms of hypoglycemia according to the Edinburgh Hypoglycemia Scale | up to 3 hours after ingestion of the liquid mixed-meal
  The Edinburgh Hypoglycemia Scale is a classification of the 11 most common symptoms of hypoglycemia. Subjective intensity-grading:
  * no symptoms 0
  * light symptoms 1
  * moderate symptoms 2
  * severe symptoms 3
Nadir plasma glucose (mmol/l) | up to 3 hours after ingestion of the liquid mixed-meal
  Nadir plasma glucose (mmol/l)
Change in proinsulin to insulin ratio in serum | at baseline and 60 min after ingestion of the mixed meal
  Change in proinsulin to insulin ratio in serum
Change in inflammatory state | at baseline and 60 min after ingestion of the mixed meal
  Change in inflammatory laboratory parameters (Interleukin (IL)1ß, IL6, Tumor necrosis factor (TNF) α, IL-10, IL-1Ra) in supernatants of Lipopolysaccharide (LPS)-stimulated and unstimulated peripheral blood mononuclear cells (PBMC)
Change in RNA sequencing (RNAseq) in peripheral PBMC | at baseline and 60 min after ingestion of the mixed meal
  Change in RNAseq in peripheral PBMC

CONTACTS AND LOCATIONS:
Overall Officials: Marc Y. Donath, Prof. Dr. med., Principal Investigator — Division of Endocrinology, Diabetes and Metabolism, University Hospital Basel
Locations (1):
- Department of Endocrinology, Diabetes and Metabolism, University Hospital Basel, Basel, Switzerland